CLINICAL TRIAL: NCT00906399
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study to Evaluate the Efficacy and Safety of PEGylated Interferon Beta-1a (BIIB017) in Subjects With Relapsing Multiple Sclerosis
Brief Title: Efficacy and Safety Study of Peginterferon Beta-1a in Participants With Relapsing Multiple Sclerosis
Acronym: ADVANCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 105MS301; 2008-006333-27 (EudraCT Number)
Record Dates: First submitted 2009-05-20; First posted 2009-05-21 (Estimated); Results first posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: interferon; injectable; MS; SC; PEGylated; Interferon beta-1a; relapsing; PEG; multiple sclerosis; subcutaneous
MeSH Terms: conditions — Recurrence; Multiple Sclerosis | interventions — peginterferon beta-1a

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo every 2 weeks for 48 weeks followed by 125 µg peginterferon beta-1a subcutaneously every 2 or 4 weeks for 48 weeks.
  Interventions: Drug: BIIB017 (peginterferon beta-1a); Drug: Placebo
- Peginterferon Beta-1a Q2W (Experimental): 125 µg peginterferon beta-1a subcutaneously every 2 weeks (Q2W) for 96 weeks.
  Interventions: Drug: BIIB017 (peginterferon beta-1a)
- Peginterferon Beta-1a Q4W (Experimental): 125 µg peginterferon beta-1a subcutaneously every 4 weeks (Q4W) for 96 weeks. Participants received a placebo injection 2 weeks after each active injection (in order to maintain the blind with Q2W arm).
  Interventions: Drug: BIIB017 (peginterferon beta-1a); Drug: Placebo

INTERVENTIONS:
Drug: BIIB017 (peginterferon beta-1a) — Supplied as a liquid in pre-filled syringes to deliver 0.5 mL of 0.25 mg/mL (125 µg dose), self-administered by subcutaneous injection.
  Other Names: PEG IFN ß-1a; PEGylated interferon beta-1a; Plegridy
Drug: Placebo — Matched placebo provided in pre-filled syringes, to deliver 0.5 mL self-administered by subcutaneous injection.
  Arms: Peginterferon Beta-1a Q4W; Placebo

SUMMARY:
The primary objective of this study is to determine the efficacy of peginterferon beta-1a in reducing the annualized relapse rate (ARR) in participants with relapsing multiple sclerosis (RMS) at 1 year. The secondary objectives of this study are to determine whether peginterferon beta-1a, at 1 year when compared with placebo, is effective in reducing the total number of new or newly enlarging T2 hyperintense lesions on brain magnetic resonance imaging (MRI) scans, reducing the proportion of participants who relapse, and slowing the progression of disability.

DETAILED DESCRIPTION:
This is a global multicenter, randomized, double-blind, parallel-group, placebo-controlled study. The treatment period is 96 weeks (2 years) in duration. Treatment Year 1 (Week 0 to Week 48) is referred to as the placebo-controlled treatment period of the study. At the beginning of Treatment Year 1, participants were randomized to receive placebo, peginterferon beta-1a 125 μg every 2 weeks, or peginterferon beta-1a 125 μg every 4 weeks. At the end of Treatment Year 1, participants in the placebo group were re-randomized to receive peginterferon beta-1a treatment so that during treatment Year 2 (Weeks 48 to Week 96) all participants received peginterferon beta-1a 125 μg every 2 or every 4 weeks. Per protocol, all primary and secondary endpoints pertain to Year 1 data.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have a confirmed diagnosis of relapsing multiple sclerosis (RMS), as defined by McDonald criteria 1 through 4 (Polman, 2005)
* Must have an EDSS score between 0.0 and 5.0.
* Must have experienced at least 2 relapses that have been medically documented within the last 3 years with at least one occurring in the last 12 months

Key Exclusion Criteria:

* Other chronic disease of immune system, malignancies, urologic, pulmonary, gastrointestinal disease
* Pregnant or nursing women
* Prior treatment with interferon could not exceed 4 weeks and subjects must have discontinued interferon treatment 6 months prior to Baseline

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1516 (Actual)
Dates: Start 2009-06; Primary Completion 2012-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (143):
- United States (12):
  - Research Site, Phoenix, Arizona
  - Research Site, Ponte Vedra Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Des Moines, Iowa
  - Research Site, Lexington, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, Teaneck, New Jersey
  - Research Site, Raleigh, North Carolina
  - Research Site, Akron, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Franklin, Tennessee
  - Research Site, Round Rock, Texas
- Belgium (2):
  - Research Site, Brussels
  - Research Site, Sint-Truiden
- Bulgaria (2):
  - Research Site, Plovdiv
  - Research Site, Sofia
- Canada (2):
  - Research Site, London, Ontario
  - Research Site, Montreal, Quebec
- Research Site, Santiago, Chile
- Colombia (3):
  - Research Site, Barranquilla, Atlántico
  - Research Site, Bogota, Cundinamarca
  - Research Site, Bogotá
- Croatia (2):
  - Research Site, Osijek
  - Research Site, Zagreb
- Czechia (7):
  - Research Site, Brno
  - Research Site, Olomouc
  - Research Site, Ostrava
  - Research Site, Ostrava - Vitkovice
  - Research Site, Ostrava-Poruba
  - Research Site, Prague
  - Research Site, Teplice
- Estonia (3):
  - Research Site, Pärnu
  - Research Site, Tallinn
  - Research Site, Tartu
- France (5):
  - Research Site, Amiens
  - Research Site, Clermont-Ferrand
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Nice
- Research Site, Tbilisi, Georgia
- Germany (15):
  - Research Site, Bayreuth
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Cologne
  - Research Site, Erbach im Odenwald
  - Research Site, Erlangen
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Leipzig
  - Research Site, Marburg
  - Research Site, München
  - Research Site, Münster
  - Research Site, Prien am Chiemsee
  - Research Site, Ulm
  - Research Site, Westerstede
- Greece (2):
  - Research Site, Athens
  - Research Site, Thessaloniki
- India (19):
  - Research Site, Ahmedabad, Gujarat
  - Research Site, Rajkot, Gujarat
  - Research Site, Bangalore, Karnataka
  - Research Site, Indore, Madhyr Pradesh
  - Research Site, Mumbai, Maharashtra
  - Research Site, Nagpur, Maharashtra
  - Research Site, Nashik, Maharashtra
  - Research Site, Pune, Maharashtra
  - Research Site, New Delhi, National Capital Territory of Delhi
  - Research Site, Saket, National Capital Territory of Delhi
  - Research Site, Amritsar, Punjab
  - Research Site, Jaipur, Rajasthan
  - Research Site, Chennai, Tamil Nadu
  - Research Site, Coimbatore, Tamil Nadu
  - Research Site, Kolkata, West Bengal
  - Research Site, Bangalore
  - Research Site, Mangalore
  - Research Site, Navi Mumbai
  - Research Site, Nehru Nagar
- Research Site, Riga, Latvia
- Mexico (5):
  - Research Site, Aquas Calientes
  - Research Site, Chihuahua City
  - Research Site, Mexico City
  - Research Site, Monterrey, Nuevo Leon
  - Research Site, Tijuana, Baja California
- Netherlands (2):
  - Research Site, Breda
  - Research Site, Nieuwegein
- New Zealand (3):
  - Research Site, Auckland
  - Research Site, Christchurch
  - Research Site, Dunedin
- Peru (2):
  - Research Site, Lima
  - Research Site, San Isidro
- Poland (15):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Gmina Końskie
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Olsztyn
  - Research Site, Plewiska
  - Research Site, Poznan
  - Research Site, Szczecin
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Zabrze
- Romania (6):
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Campulung Muscel
  - Research Site, Iași
  - Research Site, Sibiu
  - Research Site, Târgu Mureş
- Russia (12):
  - Research Site, Chelyabinsk
  - Research Site, Kaluga
  - Research Site, Kazan'
  - Research Site, Krasnodar
  - Research Site, Kursk
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Perm
  - Research Site, Rostov-on-Don
  - Research Site, Smolensk
  - Research Site, Tomsk
  - Research Site, Ufa
- Serbia (3):
  - Research Site, Belgrade
  - Research Site, Kragujevac
  - Research Site, Niš
- Spain (4):
  - Research Site, Córdoba
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Seville
- Ukraine (10):
  - Research Site, Chernivtsi
  - Research Site, Dnipropetrovsk
  - Research Site, Donetsk
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Odesa
  - Research Site, Poltava
  - Research Site, Simferopol
  - Research Site, Ternopil
  - Research Site, Vinnytsia
- United Kingdom (4):
  - Research Site, London
  - Research Site, Nottingham
  - Research Site, Salford
  - Research Site, Sheffield

REFERENCES:
- [Result] Calabresi PA, Kieseier BC, Arnold DL, Balcer LJ, Boyko A, Pelletier J, Liu S, Zhu Y, Seddighzadeh A, Hung S, Deykin A; ADVANCE Study Investigators. Pegylated interferon beta-1a for relapsing-remitting multiple sclerosis (ADVANCE): a randomised, phase 3, double-blind study. Lancet Neurol. 2014 Jul;13(7):657-65. doi: 10.1016/S1474-4422(14)70068-7. Epub 2014 Apr 30. PMID 24794721
- [Derived] Loomis SJ, Sadhu N, Fisher E, Gafson AR, Huang Y, Yang C, Hughes EE, Marshall E, Herman A, John S, Runz H, Jia X, Bhangale T, Bronson PG. Genome-wide study of longitudinal brain imaging measures of multiple sclerosis progression across six clinical trials. Sci Rep. 2023 Aug 31;13(1):14313. doi: 10.1038/s41598-023-41099-0. PMID 37652990
- [Derived] Calabresi PA, Arnold DL, Sangurdekar D, Singh CM, Altincatal A, de Moor C, Engle B, Goyal J, Deykin A, Szak S, Kieseier BC, Rudick RA, Plavina T. Temporal profile of serum neurofilament light in multiple sclerosis: Implications for patient monitoring. Mult Scler. 2021 Sep;27(10):1497-1505. doi: 10.1177/1352458520972573. Epub 2020 Dec 14. PMID 33307998
- [Derived] Cleanthous S, Cano S, Kinter E, Marquis P, Petrillo J, You X, Wakeford C, Sabatella G. Measuring the impact of multiple sclerosis: Enhancing the measurement performance of the Multiple Sclerosis Impact Scale (MSIS-29) using Rasch Measurement Theory (RMT). Mult Scler J Exp Transl Clin. 2017 Aug 15;3(3):2055217317725917. doi: 10.1177/2055217317725917. eCollection 2017 Jul-Sep. PMID 29104758
- [Derived] Scott TF, Kieseier BC, Newsome SD, Arnold DL, You X, Hung S, Sperling B. Improvement in relapse recovery with peginterferon beta-1a in patients with multiple sclerosis. Mult Scler J Exp Transl Clin. 2016 Nov 15;2:2055217316676644. doi: 10.1177/2055217316676644. eCollection 2016 Jan-Dec. PMID 28607743
- [Derived] Newsome SD, Kieseier BC, Liu S, You X, Kinter E, Hung S, Sperling B. Peginterferon beta-1a reduces disability worsening in relapsing-remitting multiple sclerosis: 2-year results from ADVANCE. Ther Adv Neurol Disord. 2017 Jan;10(1):41-50. doi: 10.1177/1756285616676065. Epub 2016 Nov 16. PMID 28450894
- [Derived] Arnold DL, Calabresi PA, Kieseier BC, Liu S, You X, Fiore D, Hung S. Peginterferon beta-1a improves MRI measures and increases the proportion of patients with no evidence of disease activity in relapsing-remitting multiple sclerosis: 2-year results from the ADVANCE randomized controlled trial. BMC Neurol. 2017 Feb 10;17(1):29. doi: 10.1186/s12883-017-0799-0. PMID 28183276
- [Derived] Newsome SD, Guo S, Altincatal A, Proskorovsky I, Kinter E, Phillips G, You X, Sabatella G. Impact of peginterferon beta-1a and disease factors on quality of life in multiple sclerosis. Mult Scler Relat Disord. 2015 Jul;4(4):350-7. doi: 10.1016/j.msard.2015.06.004. Epub 2015 Jun 14. PMID 26195056
- [Derived] Arnold DL, Calabresi PA, Kieseier BC, Sheikh SI, Deykin A, Zhu Y, Liu S, You X, Sperling B, Hung S. Effect of peginterferon beta-1a on MRI measures and achieving no evidence of disease activity: results from a randomized controlled trial in relapsing-remitting multiple sclerosis. BMC Neurol. 2014 Dec 31;14:240. doi: 10.1186/s12883-014-0240-x. PMID 25551571
- [Derived] Kieseier BC, Arnold DL, Balcer LJ, Boyko AA, Pelletier J, Liu S, Zhu Y, Seddighzadeh A, Hung S, Deykin A, Sheikh SI, Calabresi PA. Peginterferon beta-1a in multiple sclerosis: 2-year results from ADVANCE. Mult Scler. 2015 Jul;21(8):1025-35. doi: 10.1177/1352458514557986. Epub 2014 Nov 28. PMID 25432952
- [Derived] Hu X, Cui Y, White J, Zhu Y, Deykin A, Nestorov I, Hung S. Pharmacokinetics and pharmacodynamics of peginterferon beta-1a in patients with relapsing-remitting multiple sclerosis in the randomized ADVANCE study. Br J Clin Pharmacol. 2015 Mar;79(3):514-22. doi: 10.1111/bcp.12521. PMID 25265472

RESULTS

PARTICIPANT FLOW:
Groups:
- Year 1: Placebo: Placebo every 2 weeks for 48 weeks
- Year 1: Peginterferon Beta-1a Q4W; Year 2: Peginterferon Beta-1a Q4W: 125 µg peginterferon beta-1a subcutaneously every 4 weeks (Q4W) for 48 weeks. Participants received a placebo injection 2 weeks after each active injection (in order to maintain the blind with Q2W arm).
- Year 1: Peginterferon Beta-1a Q2W; Year 2: Peginterferon Beta-1a Q2W: 125 µg peginterferon beta-1a subcutaneously every 2 weeks (Q2W) for 48 weeks.
- Year 2: Placebo Followed by Peginterferon Beta-1a Q4W: Placebo every 2 weeks for 48 weeks followed by 125 µg peginterferon beta-1a subcutaneously every 4 weeks for 48 weeks. Participants received a placebo injection 2 weeks after each active injection (in order to maintain the blind with Q2W arm).
- Year 2: Placebo Followed by Peginterferon Beta-1a Q2W: Placebo every 2 weeks for 48 weeks followed by 125 µg peginterferon beta-1a subcutaneously every 2 weeks for 48 weeks.
Period: Year 1
Arm/Group | Year 1: Placebo | Year 1: Peginterferon Beta-1a Q4W | Year 1: Peginterferon Beta-1a Q2W | Year 2: Placebo Followed by Peginterferon Beta-1a Q4W | Year 2: Placebo Followed by Peginterferon Beta-1a Q2W | Year 2: Peginterferon Beta-1a Q4W | Year 2: Peginterferon Beta-1a Q2W
Started | 500 | 501 | 515 | 0 | 0 | 0 | 0
Completed Year 1 Study Treatment | 456 | 438 | 438 | 0 | 0 | 0 | 0
Completed | 456 | 438 | 439 (1 participant discontinued treatment before end of study period but remained to complete follow-up.) | 0 | 0 | 0 | 0
Not Completed | 44 | 63 | 76 | 0 | 0 | 0 | 0
Not completed — Randomized But Not Treated | 0 | 1 | 3 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 22 | 24 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 4 | 4 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 30 | 32 | 36 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 3 | 0 | 0 | 0 | 0
Not completed — Death | 2 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Other | 4 | 2 | 7 | 0 | 0 | 0 | 0
Period: Year 2
Arm/Group | Year 1: Placebo | Year 1: Peginterferon Beta-1a Q4W | Year 1: Peginterferon Beta-1a Q2W | Year 2: Placebo Followed by Peginterferon Beta-1a Q4W | Year 2: Placebo Followed by Peginterferon Beta-1a Q2W | Year 2: Peginterferon Beta-1a Q4W | Year 2: Peginterferon Beta-1a Q2W
Started | 0 | 0 | 0 | 228 | 228 | 438 | 438
Completed Year 2 Study Treatment | 0 | 0 | 0 | 200 | 196 | 391 | 411
Completed | 0 | 0 | 0 | 198 | 193 | 391 | 409
Not Completed | 0 | 0 | 0 | 30 | 35 | 47 | 29
Not completed — Adverse Event | 0 | 0 | 0 | 9 | 8 | 11 | 6
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 4 | 2 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 17 | 18 | 27 | 13
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 2 | 6 | 3
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0 | 3
Not completed — Other | 0 | 0 | 0 | 2 | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: participants who were randomized and received at least 1 dose of study treatment (peginterferon beta-1a or placebo).
Groups:
- Placebo: Placebo every 2 weeks for 48 weeks
- Peginterferon Beta-1a Q4W: 125 µg peginterferon beta-1a subcutaneously every 4 weeks (Q4W) for 48 weeks. Participants received a placebo injection 2 weeks after each active injection (in order to maintain the blind with Q2W arm).
- Peginterferon Beta-1a Q2W: 125 µg peginterferon beta-1a subcutaneously every 2 weeks (Q2W) for 48 weeks
- Total: Total of all reporting groups
Arm/Group | Placebo | Peginterferon Beta-1a Q4W | Peginterferon Beta-1a Q2W | Total
Number analyzed (Participants) | 500 | 500 | 512 | 1512
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (9.74) | 36.4 (9.87) | 36.9 (9.79) | 36.5 (9.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 358 | 352 | 361 | 1071
  Male | 142 | 148 | 151 | 441
Expanded Disability Status Scale (EDSS) [Mean (Standard Deviation); unit: units on a scale] — The EDSS measures the disability status of people with multiple sclerosis (MS) on a scale that ranges from 0 to 10. The range of main categories include 0 (normal neurologic exam), to 5 (ambulatory without aid or rest for 200 meters/disability severe enough to impair full daily activities), to 10 (death due to MS).
  units on a scale | 2.44 (1.180) | 2.48 (1.244) | 2.47 (1.255) | 2.46 (1.226)

OUTCOME MEASURES:

1. Primary Outcome: Annualized Relapse Rate (ARR) at 1 Year
Description: A relapse is defined as new or recurrent neurologic symptoms not associated with fever or infection, lasting for at least 24 hours, and accompanied by new objective neurologic findings. Only relapses confirmed by an independent neurology evaluation committee (INEC) are included in the analysis. Data after participants switched to alternative multiple sclerosis (MS) medications are excluded. Data were analyzed using negative binomial regression, adjusted for baseline Expanded Disability Status Scale (EDSS) score (< 4 versus ≥ 4), baseline age (< 40 versus ≥ 40 years), and baseline relapse rate (number of relapses in 3 years prior to study entry divided by 3).
Time Frame: 1 Year
Population: Intent-to-treat (ITT) population: participants who were randomized and received at least 1 dose of study treatment (peginterferon beta-1a or placebo).
Measure: Number (95% Confidence Interval); unit: relapses per person-years
Arm/Group | Year 1: Placebo | Year 1: Peginterferon Beta-1a Q4W | Year 1: Peginterferon Beta-1a Q2W
Number analyzed (Participants) | 500 | 500 | 512
relapses per person-years | 0.397 [0.328 to 0.481] | 0.288 [0.234 to 0.355] | 0.256 [0.206 to 0.318]
Statistical Analysis 1: Comparison: Year 1: Placebo vs Year 1: Peginterferon Beta-1a Q4W; Test type: Superiority or Other; p = 0.0114, Negative Binomial Regression; Based on negative binomial regression, with adjustment for baseline EDSS (< 4 versus ≥ 4), baseline relapse rate, age (< 40 versus ≥ 40 years); Rate Ratio = 0.725, 95% CI 2-sided [0.565 to 0.930]
Statistical Analysis 2: Comparison: Year 1: Placebo vs Year 1: Peginterferon Beta-1a Q2W; Test type: Superiority or Other; p = 0.0007, Negative Binomial Regression; Based on negative binomial regression, with adjustment for baseline EDSS (< 4 versus ≥ 4), baseline relapse rate, age (< 40 versus ≥ 40); Rate Ratio = 0.644, 95% CI 2-sided [0.500 to 0.831]

2. Secondary Outcome: Number of New Or Newly Enlarging T2 Hyperintense Lesions at 1 Year
Description: Number of new or newly enlarging T2 hyperintense lesions on brain magnetic resonance imaging (MRI) scans. Data observed after participants switched to alternative MS medications are excluded. Adjusted mean is based on negative binomial regression, adjusted for baseline number of T2 lesions.
Time Frame: 1 Year
Population: ITT population, with at least 1 post-baseline assessment. Missing data prior to alternative MS medications and visits after participants switched to alternative MS medications imputed based on previous visit data assuming the constant rate of lesion development or group mean at same visit.
Measure: Mean (95% Confidence Interval); unit: lesions
Arm/Group | Year 1: Placebo | Year 1: Peginterferon Beta-1a Q4W | Year 1: Peginterferon Beta-1a Q2W
Number analyzed (Participants) | 476 | 462 | 457
lesions | 10.9 (19.51) [9.6 to 12.5] | 7.9 (15.84) [6.9 to 9.0] | 3.6 (8.55) [3.1 to 4.2]
Statistical Analysis 1: Comparison: Year 1: Placebo vs Year 1: Peginterferon Beta-1a Q4W; Test type: Superiority or Other; p = 0.0008, Negative Binomial Regression; Lesion mean ratio (95% CI) and p-value based on negative binomial regression, adjusted for baseline number of T2 lesions; Lesion Mean Ratio = 0.72, 95% CI 2-sided [0.60 to 0.87]
Statistical Analysis 2: Comparison: Year 1: Placebo vs Year 1: Peginterferon Beta-1a Q2W; Test type: Superiority or Other; p < 0.0001, Negative Binomial Regression; [statistical method as in outcome 2, analysis 1]; Lesion Mean Ratio = 0.33, 95% CI 2-sided [0.27 to 0.40]

3. Secondary Outcome: Proportion of Participants Relapsed at 1 Year
Description: A relapse is defined as new or recurrent neurologic symptoms not associated with fever or infection, lasting for at least 24 hours, and accompanied by new objective neurologic findings. Only relapses confirmed by INEC were included in the analysis. Estimated proportion of participants relapsed is based on the Kaplan-Meier product limit method.
Time Frame: Year 1
Population: ITT population: participants who were randomized and received at least 1 dose of study treatment (peginterferon beta-1a or placebo). Participants who did not experience a relapse prior to switching to alternative MS medications or withdrew from study were censored at the time of switch/withdrawal.
Measure: Number; unit: proportion of participants
Arm/Group | Year 1: Placebo | Year 1: Peginterferon Beta-1a Q4W | Year 1: Peginterferon Beta-1a Q2W
Number analyzed (Participants) | 500 | 500 | 512
proportion of participants | 0.291 | 0.222 | 0.187
Statistical Analysis 1: Comparison: Year 1: Placebo vs Year 1: Peginterferon Beta-1a Q4W; Test type: Superiority or Other; p = 0.0200, Cox Proportion Hazards model — Based on Cox proportion hazards model, adjusted for baseline EDSS (< 4 versus ≥ 4), age (<40 versus ≥ 40 years), baseline relapse rate, and baseline Gd enhancing lesions (presence versus absence); Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.57 to 0.95]
Statistical Analysis 2: Comparison: Year 1: Placebo vs Year 1: Peginterferon Beta-1a Q2W; Test type: Superiority or Other; p = 0.0003, Cox Proportion Hazards model — [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.47 to 0.80]

4. Secondary Outcome: Estimated Proportion of Participants With Sustained Disability Progression at 1 Year
Description: Sustained disability progression is defined as: at least a 1.0 point increase on the EDSS from baseline EDSS ≥ 1.0 that is sustained for 12 weeks, or at least a 1.5 point increase on the EDSS from baseline EDSS = 0 that is sustained for 12 weeks. The EDSS measures the disability status of people with MS on a scale that ranges from 0 to 10. The range of main categories include 0 (normal neurologic examination), to 5 (ambulatory without aid or rest for 200 meters/disability severe enough to impair full daily activities), to 10 (death due to MS). Estimated proportion of participants with progression based on the Kaplan-Meier product limit method.
Time Frame: 1 Year
Population: ITT population: participants who were randomized and received at least 1 dose of study treatment (peginterferon beta-1a or placebo). Participants were censored at the time of withdrawal/switch if they withdrew from study or switched to alternative MS medication without a progression.
Measure: Number; unit: proportion of participants
Arm/Group | Year 1: Placebo | Year 1: Peginterferon Beta-1a Q4W | Year 1: Peginterferon Beta-1a Q2W
Number analyzed (Participants) | 500 | 500 | 512
proportion of participants | 0.105 | 0.068 | 0.068
Statistical Analysis 1: Comparison: Year 1: Placebo vs Year 1: Peginterferon Beta-1a Q4W; Test type: Superiority or Other; p = 0.0380, Cox Proportion Hazards model — Based on Cox Proportional Hazards model, adjusted for baseline EDSS (< 4 versus ≥ 4) and age (< 40 versus ≥ 40 years); Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.40 to 0.97]
Statistical Analysis 2: Comparison: Year 1: Placebo vs Year 1: Peginterferon Beta-1a Q2W; Test type: Superiority or Other; p = 0.0383, Cox Proportion Hazards model — Based on Cox Proportional Hazards model, adjusted for baseline EDSS (< 4 versus ≥ 4) and age (< 40 versus ≥ 40 years); Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.40 to 0.97]

ADVERSE EVENTS:
Time Frame: Screening through Week 96 (treatment period), plus 4 weeks (±5 days) follow-up
Description: One participant, randomized to placebo->Q4W, received one wrong dosing kit during Year 1, and was mistakenly distributed with one Q2W kit, therefore receiving study drug in Weeks 20 and 22 instead of placebo. For Year 1 safety tables, this participant was grouped with Q2W, and for Year 2 safety tables, this participant was grouped with Q4W.
Arm/Group | Year 1: Placebo | Year 1: Peginterferon Beta-1a Q4W | Year 1: Peginterferon Beta-1a Q2W | Year 2: Placebo Followed by Peginterferon Beta-1a Q4W | Year 2: Placebo Followed by Peginterferon Beta-1a Q2W | Year 2: Peginterferon Beta-1a Q4W | Year 2: Peginterferon Beta-1a Q2W
Serious Adverse Events (participants affected / at risk) | 76/499 | 70/500 | 55/513 | 42/227 | 36/228 | 67/439 | 39/438
Other Adverse Events (participants affected / at risk) | 378/499 | 466/500 | 472/513 | 190/227 | 206/228 | 373/439 | 367/438
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Year 1: Placebo (N=499) | Year 1: Peginterferon Beta-1a Q4W (N=500) | Year 1: Peginterferon Beta-1a Q2W (N=513) | Year 2: Placebo Followed by Peginterferon Beta-1a Q4W (N=227) | Year 2: Placebo Followed by Peginterferon Beta-1a Q2W (N=228) | Year 2: Peginterferon Beta-1a Q4W (N=439) | Year 2: Peginterferon Beta-1a Q2W (N=438)
Dengue Fever (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 0 | 1 | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 2 | 0 | 3 | 1 | 1 | 1
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 0 | 1
Septic Shock (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Acute Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Cervicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis Viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous Abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Benign Vulval Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Cervix Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anaphylactic Reaction (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Personality Disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Conversion Disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Multiple Sclerosis Relapse (Nervous system disorders) | 57 | 47 | 34 | 27 | 21 | 45 | 25
Multiple Sclerosis (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Carpal Tunnel Syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebral Ischaemia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebrovascular Insufficiency (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Monoparesis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neuritis Cranial (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neuromyelitis Optica (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Partial Seizures (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Partial Seizures With Secondary Generalization (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Uhthoff's Phenomenon (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subarachnoid Haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Retinal Detachment (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Venous Thrombosis Limb (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute Hepatic Failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bile Duct Stone (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Patellofemoral Pain Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Micturition Disorder (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abortion Incomplete (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Endometrial Hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Injection Site Reaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Irritability (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gait Disturbance (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Facial Bones Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Avulsion Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 2 | 1
Meniscus Lesion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Multiple Injuries (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Infected Skin Ulcer (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Bacterial Diarrhoea (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis Gangrenous (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Endometritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myometritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pelvic Inflammatory Disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyelonephritis Chronic (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Salpingo-Oophoritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Typhoid Fever (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral Tracheitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lip And/Or Oral Cavity Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sarcoidosis (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Basedow's Disease (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Schizophrenia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bulbar Palsy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Complex Partial Seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Extrapyramidal Disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Grand Mal Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Trigeminal Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiopulmonary Failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertensive Crisis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Shock (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Organising Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intestinal Strangulation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Drug-Induced Liver Injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatitis Toxic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Enthesopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sacroilitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cervical Dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ectropion Of Cervix (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epididymal Cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pelvic Adhesions (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Uterine Cervical Erosion (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Congenital Cystic Kidney Disease (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperpyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemoglobin Decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Year 1: Placebo (N=499) | Year 1: Peginterferon Beta-1a Q4W (N=500) | Year 1: Peginterferon Beta-1a Q2W (N=513) | Year 2: Placebo Followed by Peginterferon Beta-1a Q4W (N=227) | Year 2: Placebo Followed by Peginterferon Beta-1a Q2W (N=228) | Year 2: Peginterferon Beta-1a Q4W (N=439) | Year 2: Peginterferon Beta-1a Q2W (N=438)
Nasopharyngitis (Infections and infestations) | 77 | 69 | 54 | 22 | 17 | 45 | 47
Urinary Tract Infection (Infections and infestations) | 20 | 28 | 28 | 10 | 11 | 31 | 29
Upper Respiratory Tract Infection (Infections and infestations) | 27 | 16 | 28 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 21 | 25 | 22 | 6 | 13 | 18 | 17
Insomnia (Psychiatric disorders) | 19 | 18 | 28 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 165 | 206 | 225 | 70 | 64 | 122 | 126
Multiple Sclerosis Relapse (Nervous system disorders) | 154 | 111 | 90 | 50 | 52 | 95 | 63
Dizziness (Nervous system disorders) | 30 | 22 | 35 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 23 | 22 | 26 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 30 | 29 | 17 | 13 | 11 | 10 | 11
Vertigo (Ear and labyrinth disorders) | 43 | 32 | 27 | 9 | 11 | 17 | 14
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 31 | 26 | 34 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 28 | 26 | 21 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 31 | 43 | 45 | 9 | 14 | 16 | 27
Vomiting (Gastrointestinal disorders) | 11 | 37 | 26 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 23 | 22 | 18 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 30 | 97 | 99 | 27 | 27 | 60 | 58
Back Pain (Musculoskeletal and connective tissue disorders) | 57 | 64 | 62 | 11 | 19 | 31 | 32
Arthralgia (Musculoskeletal and connective tissue disorders) | 35 | 54 | 58 | 23 | 14 | 33 | 33
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 48 | 53 | 44 | 10 | 14 | 23 | 31
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 18 | 23 | 22 | 12 | 12 | 18 | 13
Injection Site Erythema (General disorders) | 33 | 282 | 315 | 119 | 135 | 211 | 212
Influenza Like Illness (General disorders) | 63 | 234 | 238 | 95 | 106 | 199 | 192
Pyrexia (General disorders) | 75 | 218 | 227 | 66 | 66 | 138 | 136
Chills (General disorders) | 23 | 92 | 88 | 28 | 29 | 52 | 41
Injection Site Pain (General disorders) | 15 | 67 | 78 | 25 | 25 | 32 | 45
Asthenia (General disorders) | 38 | 70 | 68 | 24 | 10 | 39 | 40
Injection Site Pruritus (General disorders) | 6 | 56 | 70 | 17 | 26 | 24 | 47
Fatigue (General disorders) | 49 | 55 | 52 | 10 | 21 | 26 | 32
Pain (General disorders) | 16 | 29 | 25 | 0 | 0 | 0 | 0
Hyperthermia (General disorders) | 5 | 26 | 22 | 0 | 0 | 0 | 0
Body Temperature Increased (Investigations) | 14 | 33 | 31 | 5 | 10 | 19 | 24
Alanine Aminotransferase Increased (Investigations) | 13 | 19 | 29 | 13 | 14 | 17 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.